CLINICAL TRIAL: NCT01357798
Title: Botulinum Toxin Type A Versus 0,9% Saline in Treatment of Cranial Allodynia in Patients With Headache
Brief Title: Botulinum Toxin Type A in Treatment of Cranial Allodynia in Patients With Headache
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federal University of Bahia (Other)
Responsible Party: PHD Ailton de Souza Melo, UFBA
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LHUFBA001
Record Dates: First submitted 2011-05-19; First posted 2011-05-23 (Estimated); Last update posted 2011-05-23 (Estimated); Status verified 2011-05

CONDITIONS: Headache; Allodynia
Keywords: Headache; Allodynia; Botulinum Toxin Type A
MeSH Terms: conditions — Headache; Hyperalgesia | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Btx-A: Active Comparator (Active Comparator): Botulinum Toxin group Will have the syringe with Botulinum toxin type A . During the study the patients will be following in the headache's clinic where the evaluator will graduate the pathologies' evolution.
  Interventions: Drug: Botulinum toxin type A
- Placebo Comparator (Placebo Comparator): 0,9% saline group Will have the syringe with 0,9% saline. During the study the patients will be following in the headache's clinic where the evaluator will graduate the pathologies' evolution .
  Interventions: Drug: 0,9% saline

INTERVENTIONS:
Drug: Botulinum toxin type A — Botulinum Toxin group Will have the syringe with Botulinum toxin type A . During the study the patients will be following in the headache's clinic where the evaluator will graduate the pathologies' evolution.
  Arms: Btx-A: Active Comparator
Drug: 0,9% saline — 0,9% saline group Will have the syringe with 0,9% saline. During the study the patients will be following in the headache's clinic where the evaluator will graduate the pathologies' evolution .
  Arms: Placebo Comparator

SUMMARY:
The objective of this study is evaluated if the Botulinum Toxin Type A is superior to 0,9% saline in treatment of cranial Allodynia in patients with headache.

Hypothesis

H(0): Botulinum Toxin Type A is not superior to 0,9% saline in treatment of cranial Allodynia in patients with headache

H (1): Botulinum Toxin Type A is superior to 0,9% saline in treatment of cranial Allodynia in patients with headache

DETAILED DESCRIPTION:
After adequation and approve from ethics committee on research involving human the selection of patients with tension headache or migraine according to The International Classification of Headache Disorders, 2nd Edition (ICHD II) will start in the Headache Clinic of Alcides Carneiro Universitary Hospital. Those selected will be oriented regarding to the study steps and potential risks of the procedures. The patients will catalog the occurrence of headache and use of analgesics for 30 days through daily headache. At the end of this month patients will be evaluated by a physician experienced in the treatment of headache to define the occurrence of pain or allodynia of the scalp. Data gathered in this consultation will be recorded in standardized questionnaires for the study. The questionnaire is divided: Patient's identification, illustration of the pain area and allodynea points, pain intensity by Visual Analogue Scale (VAS) and finally medication use will be collected in the Headache Diary.

The people are randomized with block permutation, security of equal distribution in two groups (number previous determined). One group with 0,9% saline and the other Botulinum Toxin A.

Finishing the application by the Researcher (Who doesn't know the result of randomization and the infiltrated containing). The patients will be submit to three evaluations: the first, 30 days after infiltration, with a doctor who didn't participate of the anterior steps and will analyze the pain intensity by Visual Analogue Scale (VAS), an episode of headache and use of painkiller trough Headache Diary. The Doctor will ask to the patient localize, if exist, the allodynia points. The others evolution visit will happen 60 and 90 days after application, with this same doctor using the same methods. Another professional, who doesn't know about the anterior steps of the study, will do the statics data analyze.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with tensional headache or migraine as The International Classification of Headache Disorders, 2nd Edition - ICHD II
* Patients from both sexes older than 18 years

Exclusion Criteria:

* Fill the diagnostics criteria for more than one type of primary headache as ICHD II
* Another neurological disease or systemic illness that causes headache.
* Condition that contraindicate the use of Study's Medication.
* Cognitive impairment
* Use of botulinum toxin within the last six months
* Blood, liver, or kidney disorders and pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Evaluate the allodynea's improvement following these criteria | six months
  Evaluate the allodynea's improvement following these criteria: Disappearing at least 50% infiltrated painful points.

SECONDARY OUTCOMES:
Evaluate the headache's improvement following these criteria: | six months
  Headache's episodes reduction at least 50% in the last month or pain intensity reduction by Visual Analogue Scale (VAS) in at least three points or dose's painkiller reduction at least 50%.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitário Alcides Carneiro, Campina Grande, Paraíba, Brazil